CLINICAL TRIAL: NCT04613011
Title: Effect of Double Tourniquet Technique on Width and Compressibility of Superficial Veins of Forearm
Brief Title: Effect of Double Tourniquet Technique on Ultrasonographic View of Forearm Veins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahaa Mohammed Refaie (Other)
Responsible Party: Sponsor-Investigator, Bahaa Mohammed Refaie, Lecturer of anesthesia and ICU sohag university, Sohag University
Organization: Sohag University (Other)
Other Study IDs: 1900
Record Dates: First submitted 2020-10-25; First posted 2020-11-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Superficial Forearm Veins Compressibility and Width
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — Checking vein width snd copression using US

SUMMARY:
Vein compressibility will be assessed after light pressure applied with the ultrasound probe. Vein compressibility will be graded as 3 (100% compressed), 2 (50-100 compressed), and 1 (less than 50% compressed). After baseline measurements were taken, a proximal tourniquet will be applied to mid-arm. Repeated measurements of depth, width, and compressibility will be taken one minute after the tourniquet was applied. Same measurements will be repeated again with second tourniquet applied 1 cm distal to the first tournique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18-60 years will participate in the study

Exclusion Criteria:

* patients with dialysis shunts, previous mastectomy on the examined side, fracture , skin lesion , burn or edema on the examined side

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Superficial forearm vein width and compressibility under ultrasonography | 1 minute after application of one proximal tourniquet
  Ultrasonography is used to measure forearm superficial veins width and compressibility
Superficial forearm vein width and compressibility under ultrasonography | 1 minute after application of two proximal tourniquet 1 cm apart
  Ultrasonography is used to measure forearm superficial veins width and compressibility

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa M Refaie, MD, Study Chair — Lecturer of anesthesia and ICU sohag university; Hosam eldeen M Marie, MD, Study Director — Consultant of anesthesia and ICU at Elhelal insurance hospital sohag; Mohammed A Ibrahim, MD, Principal Investigator — Lecturer of anesthesia and ICU sohag university
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided